CLINICAL TRIAL: NCT06194747
Title: Quality Improvement in Time to Treatment of Status Epilepticus
Brief Title: Improving Status Epilepticus Treatment Times
Acronym: QuITT-SE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Boston Children's Hospital (Other); Children's National Research Institute (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); UVA Children's Hospital (Other); Seattle Children's Hospital (Other); Phoenix Children's Hospital (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003386
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Status Epilepticus
Keywords: Status Epilepticus; Quality Improvement; Interventions
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Intervention Model Description: A stepped-wedge cluster randomized trial. This is a unidirectional crossover design in which clusters switch treatments at different time points, enabling statistically rigorous assessment of interventions while reducing ethical and resource limitations for quality improvement studies.
Who Masked: Participant
Masking Description: Participants will be masked as to whether the implementation bundle has been dissemination or implemented within the site they receive treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baseline phase (No Intervention): During this arm, sites will provide routine care.
- Adoption phase (Experimental): Following the dissemination visit, sites will actively work to implement the bundle of interventions.
  Interventions: Other: Quality improvement bundle
- Sustain phase (Experimental): During this arm, sites will actively work to sustain the implemented interventions and will be allowed to develop site-specific plan-do-study-act cycles in order to address site-specific key drivers with central data and methodological support.
  Interventions: Other: Quality improvement bundle and local PDSA cycles with central support
- Independent phase (Experimental): During this arm, sites will continue to sustain the implemented interventions and develop site-specific plan-do-study-act cycles in order to address site-specific key drivers without central data and methodological support.
  Interventions: Other: Quality improvement bundle and local PDSA cycles without central support

INTERVENTIONS:
Other: Quality improvement bundle — (1) standardizing BZD default to intranasal or buccal midazolam; (2) targeting initial BZD treatment within 10 minutes of seizure onset; (3) relocating and bundling all administration items needed to the hospital unit medication room; (4) utilizing basic seizure first aid in the initial patient assessment; (5) developing and implementing SE-specific EHR documentation; (6) multidisciplinary QI teams
  Arms: Adoption phase
Other: Quality improvement bundle and local PDSA cycles with central support — Sites will implement both the standard QI bundle as well as site-specific PDSA cycles with central data and methods support.
  Arms: Sustain phase
Other: Quality improvement bundle and local PDSA cycles without central support — Sites will implement both the standard QI bundle as well as site-specific PDSA cycles without central data or methods support.
  Arms: Independent phase

SUMMARY:
This is a stepped-wedge cluster randomized effectiveness-implementation hybrid study aimed at determining the effect of dissemination of a QI bundle on the time to treatment of SE among hospitalized, non-critically ill children. The primary study endpoint is to decrease the time from the SE diagnosis to treatment with the first dose of a benzodiazepine (BZD) as measured during hospitalization, which will decrease chances of morbidity and mortality.

DETAILED DESCRIPTION:
The overall study design is a stepped-wedge cluster randomized trial. A stepped-wedge is a unidirectional crossover design in which clusters switch treatments at different time points, enabling statistically rigorous assessment of interventions while reducing ethical and resource limitations for quality improvement studies.[1] Seven centers will be randomly assigned to implement the QI bundle at staggered 1-month intervals after a baseline period. Only the timing of the dissemination visit will be randomized; all sites will receive the same materials and perform the same activities (e.g. focus group, process map development, simulations).

This study is an effectiveness-implementation hybrid study. The effectiveness-implementation hybrid design is ideal for assessing both clinical interventions and implementation.17 Importantly, our interventions have strong face-validity, are evidence-based, low-risk and low-cost. For instance, the price to change BZD formulations is nominal (~$1 per dose), and other QI bundle interventions are primarily focused on frontline staff process changes. While testing the effect of the QI bundle on time to BZD treatment, we will utilize this framework and mixed methods analysis to measure implementation and identify barriers and facilitators. Thus, this proposal is of high-value, as it will provide randomized multicenter efficacy data while providing understanding for broad implementation following study end.

For the effectiveness component, we will utilize a stepped-wedge cluster randomized design. Based on our preliminary data, the intraclass correlation coefficient is estimated around 0.5, an overall sample size of 60 episodes will be adequate to achieve powers greater than 90%. A potential pitfall of the stepped wedge design is the potential confounding effects of temporal trends. We will mitigate this by tracking data at the primary site, which will be in the sustain phase throughout the study entirety. We reduce temporal effects of site enrollment (e.g., staffing changes, temporal trends in hospital admissions) by enrolling sites at different times throughout the calendar year.

The implementation component was designed utilizing the Practical, Robust Implementation and Sustainability Model (PRISM).[2] PRISM provides a scientifically rigorous and structured approach to implementation strategy development through domains focusing on (1) program, (2) external environment, (3) implementation and sustainability infrastructure and (4) recipients.[2] These elements are addressed as follows:

Program. Organizational readiness across the study sites will be critical for success. Our proposal is based on evidence derived from a successful single-center study. The QI bundle is low-cost and all interventions are currently FDA-approved. Our innovative de-implementation of time-consuming, low-value workflows (e.g. IV medication administration) will decrease care complexity in the initial stages of SE treatment. The QI bundle components are trialable, adaptable and reversible. Treatment results are immediately observable by stakeholders through individual outcomes (SE cessation) and shared measure and feedback data reports. We highlight improved outcomes and safety as organizational, caregiver, and patient priorities to achieve broad buy-in.

External Environment. Regulatory and professional organization priorities support our area of study and primary efficacy outcomes. Rapid treatment of SE has been identified as a quality measure by the AAN11, and guidelines for such care have been published by the AES.[3] Additionally, our study proposal further aligns with NAEC, which mandates a focus on rapid treatment of SE through pathway requirements across 260 hospitals. Data from our proposal will serve as a framework for accomplishing the goal of rapid SE treatment, which is inconsistently met at present.[4]

Implementation and sustainability infrastructure. Our infrastructure will utilize proven features associated with successful implementation projects.[5,6] Co-investigators experienced in working within pSERG will provide a bridge to the local QI and clinical teams, engaging stakeholders at all 3 organizational levels (frontline staff, mid-level management and senior administration). Measure and feedback will be emphasized through control chart data and implementation reports. Furthermore, the adaptable protocol allows for site-specific implementation strategies for the QI bundle as well as iterative PDSA development in the Sustain and Independent phases in order to address local drivers.

Recipients. Positive organizational characteristics are supported by LOS from senior hospital administrators and nurse managers. Furthermore, the co-investigators have previously collaborated with pSERG from their respective centers. Each site has access to data through Export, Transform, Load (ETL) data queries and EHR. The diverse demographics of patients is aided through intentional site selection and inclusion of nearly all ages of children. Importantly, our proposed interventions of performing basic seizure first aid and using non-IV forms of BZD aligns with those of patients and families in the ambulatory setting.[7]

ELIGIBILITY:
Inclusion Criteria:

* SE episode occurs in a male or female child aged between > 30 days to < 19 years
* Seizures meeting AT LEAST ONE of the following criteria:

  1. continuous clinically apparent seizure lasting greater than 5 minutes
  2. continuous clinically apparent seizure of any duration receiving BZD
  3. repeated seizures without return to neurological baseline within 5 minutes

Exclusion Criteria:

* SE episode occurs in a child with infantile spasms
* SE episode occurs in a child with electrographic-only seizures without clinical signs other than encephalopathy

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Time from the SE diagnosis to first dose of BZD | 30 days
  Time in minutes from SE diagnosis to treatment with the first dose of a benzodiazepine (BZD) as measured during hospitalization, which will decrease chances of morbidity and mortality

SECONDARY OUTCOMES:
Cost of hospitalization | 30 days
  Cost of hospitalization will be calculated as follows: cost per SE type x LOS

CONTACTS AND LOCATIONS:
Overall Officials: Adam Ostendorf, MD, Principal Investigator — Nationwide Children's Hospital and The Ohio State University
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- [Background] Feldstein AC, Glasgow RE. A practical, robust implementation and sustainability model (PRISM) for integrating research findings into practice. Jt Comm J Qual Patient Saf. 2008 Apr;34(4):228-43. doi: 10.1016/s1553-7250(08)34030-6. PMID 18468362
- [Background] Solberg LI, Brekke ML, Fazio CJ, Fowles J, Jacobsen DN, Kottke TE, Mosser G, O'Connor PJ, Ohnsorg KA, Rolnick SJ. Lessons from experienced guideline implementers: attend to many factors and use multiple strategies. Jt Comm J Qual Improv. 2000 Apr;26(4):171-88. doi: 10.1016/s1070-3241(00)26013-6. PMID 10749003
- [Background] Bradley EH, Holmboe ES, Mattera JA, Roumanis SA, Radford MJ, Krumholz HM. A qualitative study of increasing beta-blocker use after myocardial infarction: Why do some hospitals succeed? JAMA. 2001 May 23-30;285(20):2604-11. doi: 10.1001/jama.285.20.2604. PMID 11368734
- [Background] O'Hara KA. First aid for seizures: the importance of education and appropriate response. J Child Neurol. 2007 May;22(5 Suppl):30S-7S. doi: 10.1177/0883073807303066. PMID 17690085
- [Derived] Ostendorf AP, Loddenkemper T, Morgan LA, Appavu B, Farias-Moeller R, Harrar D, Press C, Abend NS, Gaillard WD, Bai S, Eisner M, McHenry L, Kroshus E, Vannatta K, Goodkin HP. Treating seizures faster: The Quality Improvement in Time to Treat Status Epilepticus (QuITT-SE) multicenter randomized stepped wedge clinical trial protocol. Contemp Clin Trials. 2025 Apr;151:107831. doi: 10.1016/j.cct.2025.107831. Epub 2025 Feb 8. PMID 39929261